CLINICAL TRIAL: NCT04959227
Title: Investigation of Anxiety, Depression and Physical Activity Level in Whirling Dervishes
Status: Enrolling by invitation | Type: Observational
Sponsor: Esra Keski̇n (Other)
Responsible Party: Sponsor-Investigator, Esra Keski̇n, RESEARCH ASSİSTANT, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: 2021-16
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Depression, Anxiety
Keywords: Anxiety Depression, physical activity
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- whirling dervish group: Beck Anxiety Inventory (min 0- max 63, As the score increases, the level of anxiety also increases.) Beck Depression Inventory (min 0- max 63, As the score increases, the level of depression also increases.) International Physical Activity Questionnaire
  Interventions: Other: Sema activity
- control group: Beck Anxiety Inventory (min 0- max 63, As the score increases, the level of anxiety also increases.) Beck Depression Inventory (min 0- max 63, As the score increases, the level of depression also increases.) International Physical Activity Questionnaire

INTERVENTIONS:
Other: Sema activity — sema activity 3 days a week for at least a year
  Groups: whirling dervish group

SUMMARY:
Sema, which means "to listen/hear" in lexical meaning, is a special physical activity performed in the form of rotating in different positions rhythmically with music.During the sema activity, although it is similar to dance therapy due to the cyclical movements it contains, it can also be evaluated as a physical activity. With Sema music therapy accompanied by musical melodies, it is similar to meditation, as the ties with the world are cut off and the attempt is made to reach divine love. Various studies have shown that physical activity, music therapy, dance therapy, and meditation have positive effects on depression and anxiety in the literature. However, there is no scientific study in the literature investigating the effects of Sema activity, which includes all these approaches, on depression, anxiety and physical activity. In order to support the literature in this sense, this study was planned to examine the effects of Sema activity on physical activity level, depression and anxiety. Individuals between the ages of 18-60 who are registered in Konya Mevlana Cultural Center who have been doing Sema for at least 1 year will be included in the study. Participants who agree to participate in the study will be asked to fill in the online Informed Volunteer Form, Demographic Information Form, Beck Anxiete Scale, Beck Depression Scale and International Physical Activity Scale - Short Form. The data will be analyzed statistically with SPSS version 23.0.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Between the ages of 18-60
* Performing Sema for at least 1 year
* Doing sema regularly (at least 3 times a week)

Exclusion Criteria:

* Being diagnosed with depression
* Having any psychiatric illness
* Presence of chronic disease (hypertension, diabetes, neurological diseases, cancer etc.)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample size of the study was calculated at a 0.90 confidence interval in line with the analyzes made with G-Power, and it was aimed to reach 30 people for each group (Leite, J.R. et al., 2010).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Depression | including last seven days- instant
  Beck Depression Inventory
Anxiety | including last seven days- instant
  Beck ANxiety Inventory
Physical Activity Level | including last seven days- instant
  International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylül Üniversitesi, Balıkesir, Turkey (Türkiye)